CLINICAL TRIAL: NCT05935527
Title: Assess the Safety, Tolerability and Efficacy of Latanoprost Liposome for Lower Eyelid Steatoblepharon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Ophthalmic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: POLAT-001-CS-402b
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-08

CONDITIONS: Lower Eyelid Steatoblepharon
Keywords: Steatoblepharon; Eyebag; Under eyelid
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, PI, sponsor will be masked until visit 5 at which time unmasking will occur to whether placebo or treatment so that placebo subjects can cross over to receive active treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Normal Saline) (Placebo Comparator): Subjects will be randomized 1:5 (1 Placebo subject to 5 receiving active treatment) to receive placebo (Normal Saline) with a volume of 120 microliters injection.
  Interventions: Drug: Placebo
- POLAT-001 (Experimental): Subjects will be randomized 1:5 (1 Placebo subject to 5 receiving active treatment) to receive POLAT-001 with a volume of 120 microliters injection, at either 1 mg/mL or 2 mg/mL
  Interventions: Drug: POLAT-001

INTERVENTIONS:
Drug: POLAT-001 — Subjects will be randomized to receive three injections per under eyebag, either 1 mg/mL or 2 mg/mL and 120 microliter volume, at each of three treatment visits.
  Arms: POLAT-001
Drug: Placebo — Subjects will be randomized to receive three injections of 120 microliters total of Normal Saline per under eyebag at each of three treatment visits.
  Other Names: Normal Saline
  Arms: Placebo (Normal Saline)

SUMMARY:
This trial is testing a drug to see if multiple injections to the undereye bags of selected patients decreases the volume of the eyebags as compared to placebo. Subjects will be randomized to receive either one of two doses of POLAT-001 or placebo. POLAT-001 will be injected into the eyebags at three of the visits. Each subject will attend 7-10 clinic visits over 98 to 140 days total to assess efficacy and safety.

DETAILED DESCRIPTION:
This trial is a proof-of-concept trial and is testing a drug to see if multiple injections to the undereye bags of selected patients decreases the volume of the eyebags as compared to placebo. Subjects will be randomized to receive either one of two doses of POLAT-001 (1 mg/mL or 2 mg/mL) or placebo (normal saline). POLAT-001 will be injected into the eyebags at three of the visits. Each subject will attend 7-10 clinic visits total over 98 to 140 days to assess efficacy and safety. Subjects assigned to placebo will crossover to receive active treatment. Efficacy will be determined using questionnaires and photography. Safety will be assessed by subject-reported events and investigator observations of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, 22 years or older with moderate to severe convexity or fullness associated with periorbital fat.
* Subject has moderate to severe eyebags per Goldberg and Simon's Orbital Fat Grading System, per protocol requirements.
* Willing and able to attend all study visits.

Exclusion Criteria:

* Any signs or symptoms of periorbital disease in the study eye and related complications, as determined by the investigator.
* Active thyroid eye disease, chronic ocular inflammatory orbital disease or other ophthalmic disease that could confound study results.
* Evidence of infection, or clinically significant periocular, periorbital or conjunctival inflammation or conditions that in the opinion of the investigator would constitute a risk or could confound the study results.
* History of hypersensitivity to prostaglandin analogs or prostaglandin PF2alpha treatments.
* Known hypersensitivity to any component of the investigational product formulation.
* Use of periocular corticosteroids within 2 months prior to Screening.
* Use of intravitreal (IVT) injections within 3 weeks prior to Screening in the study eye.
* Surgical or laser treatment of the eye or surrounding anatomical structures within 6 months prior to Screening in the study eye.
* Previous history of lower incisional eyelid surgery.
* Previous history of undereye lid tattoo or underage lash extensions.
* Previous history of infra-orbital or anterior medical cheek fillers within 24 months prior to Screening.
* The subject has received botulinum toxin treatment of the inferior pretarsal orbicularis oculi muscle within 6 months of the first injection.
* History of ocular trauma in the study eye within 6 months prior to Screening.
* Any concurrent disease that would require medical or surgical intervention during the study in the study eye (e.g., retinal detachment, significant cataract, uncontrolled glaucoma).
* Facial nerve injury or abnormal weakness, other facial rejuvenation injections (not including botulinum toxin) in the treated area, facial surgery, or facial trauma within 3 months prior to Screening. History or concurrent systemic condition that would preclude the safe administration of the study treatment or confound the results of the safety (e.g., renal or hepatic impairment).
* Any laboratory findings that based on clinical assessment of the investigator would place the subject at risk or could confound th study results.
* Significant infraorbital vascular prominence.
* Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.
* Participation in an interventional clinical study within 30 days prior to Screening.
* Any other criterion that based on the clinical judgement of the investigator may place the subject at risk or confound study results.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Mean change of photonumeric volume of eyebags in the POLAT-001 treated and placebo dose groups as measured by a 3D photography system | Baseline to 28 days after the last treatment cycle

SECONDARY OUTCOMES:
Proportion of eyebags in the POLAT-001 treated and placebo dose groups with at least 10% reduction in photonumeric volume as measured by a 3D photography system | Baseline to 28 days after the last treatment
Proportion of eyebags in the POLAT-001 treated and placebo dose groups with at least 30% reduction in photonumeric volume as measured by a 3D photography system | Baseline to 28 days after the last treatment cycle
Mean change in photonumeric volume of eyebags between the POLAT-001 treated high and low dose groups as measured by a 3D photography system | Baseline to 28 days after the last treatment cycle

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical Associates, Inc., Newport Beach, California
  - Skin Associates of South Florida, Coral Gables, Florida
  - Austin Institute for Clinical Research, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No